CLINICAL TRIAL: NCT03018535
Title: A Randomized Controlled Trial of Rituximab Versus Steroids and Cyclophosphamide in the Treatment of Idiopathic Membranous Nephropathy
Brief Title: Rituximab Versus Steroids and Cyclophosphamide in the Treatment of Idiopathic Membranous Nephropathy
Acronym: RI-CYCLO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: University of Bari (Other); Azienda Ospedaliera Brotzu (Other); University of Messina (Other); University of Milan (Other); Universita di Verona (Other); University of Chieti (Other); University of Bologna (Other); Azienda Sanitaria Locale Roma E (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Regione Piemonte (Other); University of Modena and Reggio Emilia (Other); University of Pisa (Other); University of Milano Bicocca (Other); Humanitas Hospital, Italy (Other); Azienda Ospedaliera Universitaria Policlinico (Other); Fondazione Salvatore Maugeri (Other); University of Bern (Other); University of Alberta (Other); Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Francesco Scolari, DIRECTOR OF THE DIVISION OF NEPHROLOGY, MONTICHIARI HOSPITAL, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2011 006115-59
Record Dates: First submitted 2017-01-09; First posted 2017-01-12 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Glomerulonephritis, Membranous
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Rituximab; Methylprednisolone; Methylprednisolone Hemisuccinate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RITUXIMAB (Experimental): 1 g. IV of Rituximab on days 1 and 15
  Interventions: Drug: Rituximab
- Corticosteroids and Cyclophosphamide (Active Comparator): Month 1, 3 and 5: 1g IV methylprednisolone daily for 3 doses; oral methylprednisolone (0.4mg/kg/day) or prednisone (0.5/mg/kg/day); Month 2, 4 and 6: Oral Cyclophosphamide (2.0 mg/kg/day)
  Interventions: Drug: Methylprednisolone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Rituximab — Rituximab,1 g IV, day 1 and day 15
  Other Names: Mabthera; Rituxan
  Arms: RITUXIMAB
Drug: Methylprednisolone — Methylprednisolone 1 g IV daily for 3 doses, then oral methylprednisolone (0.4 mg/kg/day) or oral prednisone (0.5mg/kg/day) for 27 days during Month 1, 3, 5.
  Other Names: URBASON; SOLUMEDROL
  Arms: Corticosteroids and Cyclophosphamide
Drug: Cyclophosphamide — Month 2, 4 and 6: Oral Cyclophosphamide (2.0 mg/kg/day) for 30 days
  Other Names: Cytoxan; Endoxan
  Arms: Corticosteroids and Cyclophosphamide

SUMMARY:
Idiopathic Membranous nephropathy (IMN) is an auto-immune glomerular disease. Recent studies suggest that circulating auto-antibodies against the podocyte surface antigens phospholipase A2 receptor1 (PLA2R1) and thrombospondin type 1 domain-containing 7A (THSD7A) cause the disease in the majority of the patients. Additional autoantibodies, directed to podocyte neo-expressed cytoplasm proteins have been described, including aldose reductase (AR), Mn-superoxide dismutase (SOD2) and alpha-enolase (alpha-ENO).

The commonest presentation of IMN is nephrotic syndrome. Data from placebo arms of interventional studies show that 30-40% of the untreated patients with persistent nephrotic syndrome (NS) progress to end-stage renal disease (ESRD).

The best-validated treatment regimen of IMN is combination therapy with steroids and cyclophosphamide, capable to induce remission of protenuria in two-third of the patients.

Despite this evidence of efficacy, there are concerns about the use of cyclophosphamide, since it may be associated with adverse events, including bone marrow suppression, gonadal toxicity, infections and oncogenic effects. Thus, the availability of alternative therapies highly effective but with a greater safety profile is desirable.

Given the key role of IgG antibodies in IMN, B cell depletion may favourably impact the glomerular disease. The anti-CD20 monoclonal antibody Rituximab is a selective B cell depleting agent. There is evidence that Rituximab is effective in the treatment of other diseases in which B cells play a key role, such as ANCA-related vasculitis. Observational studies in IMN provided encouraging data; in addition, the drug seems well tolerated.

Head-to-head comparisons between Rituximab and steroid plus ciclophosphamide in randomized clinical trials are missing.

The investigators propose this study in order to test, in a randomized controlled trial, the hypothesis that Rituximab is more effective than cyclical steroid/alkylating-agent therapy in inducing remission in patients with IMN and NS undergoing the initial treatment. In addition, the levels of the above-mentioned pathogenetic autoantibodies will be measured at baseline and during treatment. Finally, the study will compare the safety profile of steroid plus cyclophosphamide and Rituximab by evaluating the rate and severity of adverse events

DETAILED DESCRIPTION:
Idiopathic Membranous nephropathy (IMN) is an immune-mediated glomerular disease characterized by deposition of IgG4 antibodies in the subepithelial area of the glomerular basement membrane (GBM). Proteinuria is the hallmark of the disease. The commonest presentation of IMN is nephrotic syndrome with preserved kidney function. The natural course of the disease can be variable and may be punctuated with spontaneous remissions and relapses. In about 20% of patients, there is spontaneous complete remission of the nephrotic syndrome, and another 15-20% undergo partial remission; about 30% of patients may remain with fluctuating proteinuria and about 30% may progress to end-stage renal disease (ESRD). However, data from natural history studies and placebo arms of intervention studies with follow-up lasting more than 10 years show that about 30-40% of the untreated patients with persistent nephrotic syndrome progress to ESRD.

Complete remission of nephrotic syndrome predicts excellent long-term kidney and patient survival, and partial remission also significantly reduces the risk of progression to ESRD. Therefore, persisting remission of the nephrotic state is an acceptable surrogate end-point to assess efficacy of treatment. The primary aims of treatment, therefore, are to induce a lasting reduction in proteinuria. The best-validated regimen is combination therapy with corticosteroids and cyclophosphamide ("Ponticelli" regimen). This treatment is superior to supportive therapy alone in inducing remissions and preventing long-term decline of kidney function in patients with idiopathic MN and persisting nephrotic syndrome. However, there are concerns about the use of cyclophosphamide, since its use may be associated with adverse events, leading to treatment interruption in about 9% of patients. These adverse events include bone marrow suppression, gonadal toxicity, infections and oncogenic effects.

Thus, the availability of alternative therapies highly effective but with a greater safety profile is desirable.

Recent human studies confirmed that MN is an autoimmune disease, suggesting that the disease may be triggered by isotype specific autoantibodies directed against podocyte enzymes and podocyte receptors that are recognized as antigens, including M-type phospholipase-2 receptors(PLA2R1) and thrombospondin type 1 domain-containing 7A (THSD7A). The podocyte expression of these autoantigens can trigger the production of specific antibodies and in situ deposits of immune complexes, with consequent activation of complement cascade, oxygen radicals, and other inflammatory pathways leading to tissue injury and fibrosis. Additional autoantibodies, directed to podocyte neo-expressed cytoplasm proteins have been described, including aldose reductase (AR), Mn-superoxide dismutase (SOD2) and alpha-enolase (alpha-ENO).

However, the mechanisms eliciting the expression of these neoantigens on podocytes and regulating the deposition of the auto-antibodies on the subepithelial surface of the glomerular basement membrane is not known.

Considering the potential role of IgG antibodies in the pathogenesis of IMN, B cell depletion may favourably impact the glomerular disease as reflected by a reduction in proteinuria. The anti-CD20 monoclonal antibody Rituximab is a selective B cell depleting agent, capable to maintain B cells undetectable for 3-12 months. There is evidence that this strategy is effective in the treatment of other diseases in which B cells play a key role, such as ANCA-related vasculitis and humoral allograft rejection. Preliminary studies in IMN are promising, with observational studies providing encouraging data; in addition, the drug seems well tolerated with minimal adverse events.

Head-to-head comparisons between Rituximab and steroid plus ciclophosphamide in randomized clinical trials are missing.

The investigators propose this study in order to test in a randomized controlled trial the hypothesis that selective B lymphocyte depletion obtained with Rituximab is more effective than cyclical corticosteroid/alkylating-agent therapy in inducing long-term remission of proteinuria in patients undergoing the initial treatment of with IMN and nephrotic syndrome. In addition, since specific assay for the above-mentioned autoantibodies are now available, the levels of these pathogenetic autoantibodies will be measured at baseline and during treatment. Finally, the study will compare the safety profile of steroid plus cyclophosphamide and Rituximab by evaluating the rate and severity of adverse events.

Design and Power Considerations

The investigators hypothesized that the remission probability in the RTX arm will be greater than in the active comparator group (superiority design). Available data (Ponticelli 1998) suggest that the probability of complete remission with standard therapy is 15% at one year.

The investigators plan to enroll 70 patients in this pilot RCT. This sample size will be able to detect with a power of 80% (and a two-sided P of 0.05) an odds ratio of 3, i.e. change in probability from 0.15 to 0.45 - a very optimistic effect. Smaller (and likely more reasonable) effects would require larger studies.

The study will provide an estimate of this true effect, if it exists.

Adverse effects:

Patients will be directly questioned every two weeks during the drug exposure and then at monthly intervals during follow-up. In addition a contact number will be provided to the subjects to call if they experience any adverse affect or if they suspect adverse effect at any time between specific visits

Definition Of Proteinuric Status

UP = urinary protein (g/24h)

Complete remission (CR) UP ≤ 0.3 g

Partial remission (PR): Reduction in UP of > 50% plus final UP ≤ 3.5 g but >0.3g

Non-response (NR): Reduction in UP of < 50% (includes increase in UP <50%)

Neither CR nor PR

Progression: Proteinuria /S. creatinine increases by > 50% over the baseline

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven diagnosis of idiopathic MN performed within the past 24 months
2. Proteinuria > 3.5 g/24h on three 24-hour urine collection (once a week for 3 weeks)
3. Estimated GFR (MDRD formula) ≥ 30ml/min/1.73m2 under ACEI/ARB therapy
4. Post-menopausal females, or females surgically sterile or practicing a medically approved method of contraception (no birth-control pill)
5. Three months of ACEI and/or ARB therapy before treatment
6. Blood Pressure <130/80 mm Hg
7. HMG-CoA reductase inhibitor therapy
8. Patients remaining with proteinuria >3.5g/24h after 3 months of ACEI and/or ARB therapy and Blood Pressure <130/80 mm Hg may be randomized to RTX / cyclical corticosteroid/alkylating-agent therapy without the need of the run-in/conservative phase of the study.

Exclusion Criteria:

1. serum creatinine >2.5 mg/dl; Estimated GFR < 30 ml/min/1.73m2
2. previous treatment with Rituximab, Steroids, Alkylating Agents, Calcineurin Inhibitors, Synthetic ACTH, MMF, Azathioprine
3. Presence of active infection
4. Secondary cause of MN (e.g. hepatitis B, SLE, medications, malignancies). Testing for HIV, Hepatitis B and C should have occurred < 6 months prior to enrollment into the study
5. Type 1 or 2 diabetes mellitus
6. Pregnancy or nursing for safety reasons
7. Renal vein thrombosis documented prior to entry by renal US or CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
change in probability of complete remission (proteinuria < 0.3 g/day) Primary Outcome Measures The primary outcome measure is the change in probability of complete remission (proteinuria < 0.3 g/day) at one year (see Design and power considerations). | 1 year
  The primary outcome measure is the change in probability of complete remission (proteinuria < 0.3 g/day) at one year

SECONDARY OUTCOMES:
Change from baseline in proteinuria | from randomization up to 36 months
  Change from baseline in proteinuria at 6,12, 18, 24 and 36 months following treatment
CR (Complete Remission) or PR (Partial Remission: Reduction in UP of > 50% plus final UP ≤ 3.5 g but >0.3g ) | from randomization up to 36 months
  CR (Complete Remission) or PR (Partial Remission) at 6, 12, 18, 24, and 36 months
Estimated Glomerular filtration rate (MDRD formula) | from randomization up to 36 months
  Estimated Glomerular filtration rate (MDRD formula) at 6, 12, 18, 24, and 36 months
Serum creatinine level (mg/dl) | from randomization up to 36 months
  Serum creatinine level (mg/dl) at 6, 12, 18, 24, and 36 months
Frequency of and time to relapse of nephrotic syndrome | up to 36 months
  Frequency of and time to relapse of nephrotic syndrome
Frequency of auto-antibodies and its relation to therapy and proteinuria response in a subgroup of patients | baseline and after treatment (day 3, month 1, 3, 6 , 6 and 12)
  Frequency of auto-antibodies and its relation to therapy and proteinuria response in a subgroup of patients at baseline and 3 days, 1 month, 3 months, 6 months and 12 months after treatment
serious side effects: Death, Life-threatening event, Hospitalization, Disability in the patient's body function/structure or physical activity or quality of life, Congenital anomaly, Intervention to prevent permanent impairment or damage) | up to 36 months
  serious side effects: Death, Life-threatening event, Hospitalization, Disability in the patient's body function/structure or physical activity or quality of life, Congenital anomaly, Intervention to prevent permanent impairment or damage.

CONTACTS AND LOCATIONS:
Overall Officials: FRANCESCO SCOLARI, MD, Principal Investigator — Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Locations (1):
- Division of Nephrology, Montichiari Hospital, ASST Spedali Civili di Brescia, Montichiari, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glassock RJ. The pathogenesis of membranous nephropathy: evolution and revolution. Curr Opin Nephrol Hypertens. 2012 May;21(3):235-42. doi: 10.1097/MNH.0b013e3283522ea8. PMID 22388552
- [Background] Cravedi P, Remuzzi G, Ruggenenti P. Rituximab in primary membranous nephropathy: first-line therapy, why not? Nephron Clin Pract. 2014;128(3-4):261-9. doi: 10.1159/000368589. Epub 2014 Nov 22. PMID 25427622
- [Background] Murtas C, Bruschi M, Candiano G, Moroni G, Magistroni R, Magnano A, Bruno F, Radice A, Furci L, Argentiero L, Carnevali ML, Messa P, Scolari F, Sinico RA, Gesualdo L, Fervenza FC, Allegri L, Ravani P, Ghiggeri GM. Coexistence of different circulating anti-podocyte antibodies in membranous nephropathy. Clin J Am Soc Nephrol. 2012 Sep;7(9):1394-400. doi: 10.2215/CJN.02170312. Epub 2012 Jul 5. PMID 22773590
- [Background] Ponticelli C, Zucchelli P, Passerini P, Cesana B, Locatelli F, Pasquali S, Sasdelli M, Redaelli B, Grassi C, Pozzi C, et al. A 10-year follow-up of a randomized study with methylprednisolone and chlorambucil in membranous nephropathy. Kidney Int. 1995 Nov;48(5):1600-4. doi: 10.1038/ki.1995.453. PMID 8544420
- [Background] Jha V, Ganguli A, Saha TK, Kohli HS, Sud K, Gupta KL, Joshi K, Sakhuja V. A randomized, controlled trial of steroids and cyclophosphamide in adults with nephrotic syndrome caused by idiopathic membranous nephropathy. J Am Soc Nephrol. 2007 Jun;18(6):1899-904. doi: 10.1681/ASN.2007020166. Epub 2007 May 9. PMID 17494881
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952
- [Derived] Scolari F, Delbarba E, Santoro D, Gesualdo L, Pani A, Dallera N, Mani LY, Santostefano M, Feriozzi S, Quaglia M, Boscutti G, Ferrantelli A, Marcantoni C, Passerini P, Magistroni R, Alberici F, Ghiggeri GM, Ponticelli C, Ravani P; RI-CYCLO Investigators. Rituximab or Cyclophosphamide in the Treatment of Membranous Nephropathy: The RI-CYCLO Randomized Trial. J Am Soc Nephrol. 2021 Apr;32(4):972-982. doi: 10.1681/ASN.2020071091. Epub 2021 Mar 1. PMID 33649098
- [Derived] Scolari F, Dallera N, Gesualdo L, Santoro D, Pani A, Santostefano M, Feriozzi S, Mani LY, Boscutti G, Messa P, Magistroni R, Quaglia M, Ponticelli C, Ravani P. Rituximab versus steroids and cyclophosphamide for the treatment of primary membranous nephropathy: protocol of a pilot randomised controlled trial. BMJ Open. 2019 Dec 4;9(12):e029232. doi: 10.1136/bmjopen-2019-029232. PMID 31806605